CLINICAL TRIAL: NCT06189898
Title: Functional Imaging to Identify Radiosensitive Esophageal Cancer - a Biomarker Validation Study
Acronym: FIRASE
Status: Recruiting | Type: Observational
Sponsor: Sebastian Zschaeck (Other)
Collaborators: Helmholtz Zentrum Dresden Rossendorf, Dresden, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Sebastian Zschaeck, MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: FIRASE
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor biopsies and primary cell culture, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Re Staging FDG-PET — Additional interim FDG-PET during week four of preoperative or definitive chemoradiation for esophageal carcinomas. Evaluation of standardized uptake ratio (SUR) and increased uptake of non tumor affected esophagus (Delta NTO).
  Other Names: [18F]Fluorodeoxyglucose positron emission tomograhpy at week four radiochemotherapy

SUMMARY:
This trial on biomarker validation investigates the use of innovative re-staging FDG-PET parameters to detect highly chemoradiation (CRT) sensitive squamous cell carcinomas of the esophagus (SCEC) at the end of preoperative or definitive CRT.

DETAILED DESCRIPTION:
This trial on biomarker validation investigates the use of innovative re-staging FDG-PET parameters to detect highly chemoradiation (CRT) sensitive squamous cell carcinomas of the esophagus (SCEC) at the end of preoperative or definitive CRT. Successful validation of this biomarker could lead to a more individualized approach for patients, i.e. organ preservation in highly chemoradiosensitive patients. Since favorable response to CRT is associated with better outcome of patients, the primary endpoint of the study is an improved event-free-survival (EFS) in responders receiving definitive CRT compared to non-responders. Additional quality of life and other important endpoints (side effects, overall survival, local control, occurrence of distant metastases) will be assessed in both treatment groups.

The investigated PET parameters are Maximum standardized uptake ratio (SURmax) of the primary tumor at week four of chemoradiation and change of maximum standardized uptake value of the non tumor affected esophagus (DeltaNTO).

To improve the treatment in non-responders in future trials, the study has two additional scientific support programmes included: Genetic sequencing of tumor tissue to identify targetable mutations and correlate these with novel imaging biomarkers of none-response on the one hand (biology based treatment optimization). On the other hand the study will include an additional observational study arm. In this arm patients with adenocarcinoma of the esophagus can be included. Our biomarker has only been established in squamous cell carcinomas, therefore it is an interesting exploratory question, if the parameter can also be applied to patients with adenocarcinomas of the esophagus. An additional scientific support program will establish primary tumor cells for better mechanistical understanding of the imaging biomarkers and testing of treatment according to targetable mutations.

ELIGIBILITY:
Inclusion Criteria:

* patients with squamous cell, undifferentiated or adenocarcinoma of the esophagus, UICC stage II-IVA (maximum T4a)
* ECOG performace status 0-2
* Complete clinical staging, including, esophagogastroscopy, EUS, CT neck/thorax/abdomen and adequate pulmonary function.
* Adequate hematological, renal, hepatic and pulmonary functions defined as:

granulocytes ≥ 1.5 x 109/l platelets ≥ 100 x 109/l total bilirubin ≤ 1.5 x upper normal limit creatinine ≤ 120 μmol/L FEV1 ≥ 1.5 L

* Written, voluntary informed consent
* Willingness to perform effective contraceptive practices during treatment for patients with childbearing potential

Exclusion Criteria:

* Evidence of distant metastases (cM1)
* Prior high-dose radiotherapy to the thorax or abdomen
* Primary tumor cT4b
* history or concurrent malignancy as judged by the treating physician. This is only an exclusion criterion if the other malignancy is considered the oncological potentially leading cause of death compared to the esophageal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the primary endpoint only patients with squamous cell histology will be evaluated. Patients with adenocarcinomas will be used as exploratory cohort.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | continiously with two year follow up
  progression free survival is defined as any tumor recurrence (local, regional and or distant) or death

SECONDARY OUTCOMES:
Overall survival | continiously with two year follow up
  death of patients
loco-regional recurrence free survival | continiously with two year follow up
  time without local or regional tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Zschaeck, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zschaeck S, Li Y, Butof R, Lili C, Hua W, Troost ECG, Beck M, Amthauer H, Kaul D, Kotzerke J, Baur ADJ, Ghadjar P, Baumann M, Krause M, Hofheinz F. Combined tumor plus nontumor interim FDG-PET parameters are prognostic for response to chemoradiation in squamous cell esophageal cancer. Int J Cancer. 2020 Sep 1;147(5):1427-1436. doi: 10.1002/ijc.32897. Epub 2020 Feb 19. PMID 32010957